CLINICAL TRIAL: NCT06456450
Title: Taiwan Severe Asthma Biologic Registry
Acronym: TARGET
Status: Recruiting | Type: Observational
Sponsor: Taichung Veterans General Hospital (Other)
Collaborators: E-DA Hospital (Other); National Cheng-Kung University Hospital (Other); National Yang Ming Chiao Tung University Hospital (Other); Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Pin-Kuei Fu, MD, PhD, Director of Clinical Trail Center, Taichung Veterans General Hospital
Other Study IDs: CE24049B
Record Dates: First submitted 2024-05-30; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Pulmonary Disease; Asthma
Keywords: Severe Asthma; Registry; Biologic
MeSH Terms: conditions — Lung Diseases; Asthma | interventions — Omalizumab; mepolizumab; benralizumab; tezepelumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Omalizumab: Severe asthma patients who are treated with omalizumab after January 1, 2020.
  Interventions: Biological: Biological Treatment for severe asthma patients
- Mepolizumab: Severe asthma patients who are treated with mepolizumab after January 1, 2020.
  Interventions: Biological: Biological Treatment for severe asthma patients
- Benralizumab: Severe asthma patients who are treated with benralizumab after January 1, 2020.
  Interventions: Biological: Biological Treatment for severe asthma patients
- Dupilzumab: Severe asthma patients who are treated with dupilzumab after January 1, 2020.
  Interventions: Biological: Biological Treatment for severe asthma patients
- Tezepelumab: Severe asthma patients who are treated with Tezepelumab after January 1, 2020.
  Interventions: Biological: Biological Treatment for severe asthma patients

INTERVENTIONS:
Biological: Biological Treatment for severe asthma patients — Biological treatment for severe asthma available in Taiwan and is covered by covered by National Health Insurance
  Other Names: Omalizumab; Mepolizumab; Benralizumab; Dupilzumab; Tezepelumab

SUMMARY:
This is a prospective multi-centers cohort study for registration adult patients with severe asthma and were reimbursed biologics treatment in Taiwan.

The goal of this observational study is to discover the real-world effectiveness, the impact of initiating, switching of biologics, and the possible prediction factors for selecting the best treatment option for patients.

The main question[s] it aims to answer are:

1. Determine risk factors associated with poor asthma control.
2. Support the development of effectiveness and safety of therapeutic principles
3. To discover the real-world effectiveness of different biologics ( Clinical remission)
4. To discover the impact of initiating biologics for severe asthma patients.
5. To evaluate the prevalence of biologics switching and its benefits for patients.
6. To compare the achievement rate of clinical remission among different biologics.

Participants who are treated either with omalizumab, mepolizumab, benralizumab dupilzumab or Tezepelumab after January 1, 2020 will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures.
* Patient should be reviewed as well as confirmed by the National Health Insurance Administration (NHIA) or by the study board member as a Severe Asthma case.
* Female and male aged over 18 years old.
* Patients who are treated either with omalizumab, mepolizumab, or benralizumab after January 1, 2020.

Exclusion Criteria:

* Lack of informed consent for participation.
* History of Biologic usage before January 1, 2020, should be ruled out.
* The washout period should be at least 12 months. In other words, the enrolled patients should have no experience in receiving a biological treatment or in participating relative clinical trial before his/her biologic initiation.
* Comorbid pulmonary diseases (e.g.: Chronic Obstructive Pulmonary Disease, Bronchiectasis, Pulmonary Fibrosis, etc.) or risk factors (e.g.: smoking or environmental exposure, etc..) that could be associated with pulmonary or systemic diseases, other than Asthma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Severe Asthma Patient
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-11-11 (Actual); Primary Completion 2043-02-28 (Estimated); Study Completion 2043-02-28 (Estimated)

PRIMARY OUTCOMES:
Status of Asthma Control | 6 months
  Mean change in Asthma Control Test score after biologic initiation.
Status of Asthma exacerbations | 6 months
  Annual frequency of exacerbations after biologic initiation.
Reduction of daily oral corticosteriod dose | 6 months
  Percentage of daily oral corticosteroids dose reduction after biologic initiation.
Change of Pre-BD FEV1 (%pred) | 6 months
  Measure the change of Pre-BD FEV1 (%pred) after biologic initiation. FVC (L) FEV1(L)

SECONDARY OUTCOMES:
Disease Prognosis | 6 months
  1. Describe the Cross-sectional phenotypic or pathophysiological (endotype) characteristics of poor asthma control.
  2. Describe the natural history, intervention responsiveness and long-term prognosis of severe asthma.
Mortality | 6 months
  Define the mortality rate of the study cohort

CONTACTS AND LOCATIONS:
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided